CLINICAL TRIAL: NCT04903899
Title: A Phase II Trial of 177Lutetium-DOTATATE in Children With Primary Refractory or Relapsed High-risk Neuroblastoma
Brief Title: 177Lutetium-DOTATATE in Children With Primary Refractory or Relapsed High-risk Neuroblastoma
Acronym: LuDO-N
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jakob Stenman (Other)
Collaborators: Advanced Accelerator Applications (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Jakob Stenman, Consultant Pediatric Surgeon, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuDO-N
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Neuroblastoma Recurrent; Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-DOTATATE (Experimental): A total of two doses of 177Lu-DOTATATE will be administered intravenously. The minimum time between treatments is 2 weeks.
  Interventions: Combination Product: 177Lu-DOTATATE

INTERVENTIONS:
Combination Product: 177Lu-DOTATATE — A weight-based activity of 200 MBq kg-1 will be used for the first dose. The activity of the second dose will be calculated based on whole body activity scans as well as SPECT CT scans to determine the absorbed kidney dose. The aim is to administer 177Lu-DOTATATE corresponding to a whole-body dose of 1,2 Gy, with a cumulative whole-body dose of about 2,4 Gy over two courses, and not exceeding a cumulative renal dose of 23 Gy, in order to avoid renal toxicity.

SUMMARY:
The LuDO-N Trial is a multi-centre phase II clinical trial on 177Lu-DOTATATE treatment of recurrent or relapsed high-risk neuroblastoma in children. The LuDO-N Trial builds on the experience from the previous LuDO Trial and utilises an intensified dosing schedule to deliver 2 doses over a 2-week period, in order to achieve a maximal effect on the often rapidly progressing disease. This strategy requires a readiness for autologous stem cell transplantation in all patients, but is not anticipated to increase the risk of long-term sequelae, since the cumulative radiation dose remains unchanged. The primary aim of the study is to assess the response to 177Lu-DOTATATE treatment at 1 and 4 months after ende of treatment. Secondary aims are to assess survival and treatment-related toxicity. Additional aim are to correlate tumour dosimetry with response, correlate SSTR-2 expression with 68Ga-DOTATATE uptake and to correlate the uptake with the treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology 1.1. Histologically confirmed diagnosis of neuroblastoma 1.2. Immunohistochemical staining for somatostatin receptors (SSTR) performed from primary tumor tissue when available
2. Relapsed or primary refractory high-risk neuroblastoma: INSS stage 4 disease or INRGSS stage M disease
3. Age >18 months at the time of enrolment into this study
4. Life expectancy of greater than 3 months
5. Performance Status 5.1. Karnofsky > 50% (for patients > 12 years of age) 5.2. Lansky > 50% (for patients ≤ 12 years of age)
6. Prior treatment 6.1. Two-week washout from any prior treatment 6.2. Patients must have recovery of hematological toxicity following previous therapy 6.3. Adequate recovery from major surgery prior to receiving study treatment
7. Diagnostic imaging 7.1. Uptake in the primary tumor or metastatic tumour deposits on 68Ga-DOTATATE PET/CT at least higher than the liver uptake and performed within two months prior to registration 7.2. 123I-mIBG scintigraphy to be performed within two months prior to registration 7.3. CT or MRI of the primary tumor and bulky metastatic sites within two months prior to registration
8. Laboratory requirements to be performed within 7 days prior to commencing trial treatment 8.1. Hematology: 8.1.1. Hemoglobin, If Hb is <120 g/L then patient will receive a blood transfusion prior to commencing trial treatment 8.1.2. Absolute neutrophil count > 1.0 x 109/L 8.1.3. Absolute Platelets > 50 x 109/L 8.2. Biochemistry: 8.2.1. Bilirubin within 1.5 x ULN 8.2.2. ALT within 2.5 x ULN 8.2.3. AST within 2.5 x ULN 8.2.4. GGT within 5 x ULN 8.2.5. ALP within 5 x ULN 8.2.6. Glomerular filtration rate >50mL/min/1.73m2 assessed by a recognised method, such as inulin, 51Cr-EDTA, 99mTc-DTPA or iohexol clearance and performed within 2 months prior to registration 8.2.7. Urinary catecholamine metabolites measured within 2 months prior to registration
9. Peripheral blood stem cells (PBSC) 9.1. A minimum of 2 x106 CD34+ cells/kg (optimally 6 x106 CD34+ cells/kg) must be available for each study subject prior to registration
10. Written informed consent from patient and/or parent(s) or legal guardian(s) in accordance with national regulations, prior to registration or any trial-related screening procedures

Exclusion Criteria:

1. Not fit enough to undergo proposed study treatment, as assessed by national PI, considering precautions defined in the latest version of the 177Lutetium-DOTATATE SmPC.
2. Pregnant or lactating patient
3. Concurrent treatment with any anti-tumor agents
4. Prior treatment with other radiolabeled somatostatin analogues
5. Hypersensitivity to any component of the investigational drug 177Lutetium-DOTATATE
6. Treatment with long-acting somatostatin analogues within 30 days, or with short-acting somatostatin analogues within 24 hours prior the administration of 177Lutetium-DOTATATE

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2031-05-20 (Estimated)

PRIMARY OUTCOMES:
Treatment response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC) - 1 months after End of Treatment | 1 months following end of treatment
  Treatment response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC)

SECONDARY OUTCOMES:
Number and severity of treatment-related adverse events | Up to 5 years after end of treatment
  Number and severity of treatment-related adverse events
Treatment response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC) - 4 months after End of Treatment | 4 months following end of treatment
  Treatment response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC)
Progression-free survival | Time from registration to progression or death, up to 5 years following end of treatment
  Time to progress or death, whichever occurs first
Overall survival - up to 5 years after End of Treatment | Time from registration to the the date of death, up to 5 years following end of treatment
  Overall survival

OTHER OUTCOMES:
Tumour dosimetry: absorbed dose per administration of 177Lu-DOTATATE | At every administered dose of 177Lu-DOTATATE throughout the trial treatment phase (5 years)
  Measured by SPECT/CT
Correlation of expression of Somatostatin Receptor-2 (SSTR-2) to uptake on 68Ga-DOTATOC PET/CT | Throughout the trial treatment phase (5 years)
  SSTR-2 expression in the histology samples from primary surgery measured by immunohistochemistry.
Uptake on 68Ga-DOTATOC PET/CT | At end of treatment, and 1 and 4 months after end of treatment.
  Measured by SUVmax (maximum standardized uptake value)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stenman, MD PhD, Study Chair — Karolinska University Hospital
Locations (5):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark
- Vilnius University Hospital, Vilnius, Vilnius County, Lithuania
- Princess Maxima Center for Pediatric Oncology, Utrecht, Utrecht, Netherlands
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sundquist F, Georgantzi K, Jarvis KB, Brok J, Koskenvuo M, Rascon J, van Noesel M, Gryback P, Nilsson J, Braat A, Sundin M, Wessman S, Herold N, Hjorth L, Kogner P, Granberg D, Gaze M, Stenman J. A Phase II Trial of a Personalized, Dose-Intense Administration Schedule of 177Lutetium-DOTATATE in Children With Primary Refractory or Relapsed High-Risk Neuroblastoma-LuDO-N. Front Pediatr. 2022 Mar 10;10:836230. doi: 10.3389/fped.2022.836230. eCollection 2022. PMID 35359899